CLINICAL TRIAL: NCT03629158
Title: Brief Behavioral Health Intervention Program for Patients With Stable Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Chelsea Wiener, MS, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBE-18-14085
Record Dates: First submitted 2018-07-31; First posted 2018-08-14 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease; Coronary Heart Disease
Keywords: Behavioral Medicine; Clinical Trial; Cardiology; Health Behavior; Healthy Lifestyle; Self Efficacy
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLIMB intervention (Experimental): The intervention group will receive the Cardiac Lifestyle Intervention for Maintaining healthy Behaviors ("CLIMB") intervention. Participants will participate in a 3-session, one-on-one intervention that takes place over the course of two weeks.
  Interventions: Behavioral: CLIMB intervention
- Treatment as usual (TAU) (No Intervention): The TAU group will continue to receive their regular medical care.

INTERVENTIONS:
Behavioral: CLIMB intervention — The intervention group will receive the Cardiac Lifestyle Intervention for Maintaining healthy Behaviors ("CLIMB") intervention. Participants will participate in a 3-session, one-on-one intervention that takes place over the course of two weeks. Sessions range from 1-2 hours in length, including questionnaire completion. Participants will be given information and taught relevant skills to increase engagement in lifestyle behaviors relevant to cardiac health.
  Arms: CLIMB intervention

SUMMARY:
The purpose of this study is to examine the effectiveness of a lifestyle intervention for patients living with stable coronary artery disease (CAD). One group will receive the the intervention, and the other will receive treatment as usual (TAU). The investigators hypothesize that, compared to the TAU group, participants receiving the intervention will 1) experience greater confidence in managing their cardiac disease, as indicated by perceived self-efficacy and illness perceptions; 2) experience greater psychological adjustment as indicated by depressive, anxious, and demoralization symptoms; 3) experience greater engagement in health behaviors including healthy eating and physical activity.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of two research groups: the intervention group (IG) and the treatment as usual (TAU) group. The IG will receive the Cardiac Lifestyle Intervention for Maintaining healthy Behaviors ("CLIMB"). CLIMB is a 3-session (2-week) intervention. One session includes health behavior feedback, and patient selection of relevant lifestyle modules based on values clarification. In the remaining two sessions, participants will complete two of five elective lifestyle modules: Healthy Eating, Physical Activity, Reducing Stress and Worry, Mood Management, and Smoking Cessation Education. Intervention components include information provision, goal setting, problem solving, and elements of cognitive behavioral therapy.

Participants in the IG will complete a Baseline assessment, three intervention sessions, a 30-day follow-up, and a 3-month follow-up. Baseline and Session 1 will take place on the same day. Sessions 1, 2, and 3 will be spaced approximately one week apart from one another (1 week in-between Sessions 1 and 2, and 1 week in-between Sessions 2 and 3). The 30-day follow-up will occur approximately 30-days after Session 3. The 3-month follow-up will occur approximately 3 months after Session 3. Assessment measures will be filled out at Baseline, at Post-treatment (end of Session 3), at 30-day follow-up, and at 3-month follow-up. The TAU group will fill out assessment measures at comparable time points, with the exception that there will be no 3-month follow-up. After completing their 30-day follow-up measures, TAU members may elect to receive the CLIMB intervention.

ELIGIBILITY:
Inclusion Criteria:

1. CAD as indicated by history of at least one myocardial infarction, at least one coronary artery bypass graft surgery, at least one coronary stent, and/or at least one coronary vessel with stenosis greater than or equal to 70%.
2. Stable status as indicated by no myocardial infarctions, unstable angina, or other acute coronary syndromes within the past 3 months, no coronary revascularizations within the past 3 months, and no planned revascularizations.

Exclusion Criteria:

1. Age < 30 years or > 79 years
2. Cognitive impairment as indicated by diagnosis in medical chart
3. Psychotic symptoms as indicated by diagnosis in medical chart
4. Any documented non-skin malignancy, malignant melanoma, or advanced kidney disease (indicated by stage 4 or 5 or on dialysis)
5. Ejection fraction < 30%
6. Physician determination of inappropriateness for study, due to anticipated life expectancy of <1 year, presence of a survival limiting or uncontrolled illness, and/or hemodynamically important valvular disease.
7. Women who are pregnant or breast feeding
8. Non-English-speaking
9. Participation in another clinical trial concurrently or within 30 days before screening
10. Psychological safety concerns, including plans to harm oneself within the past two months and/or suicide attempt within the past year

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Self-efficacy for managing coronary artery disease | 2-weeks/post-treatment
  Participants will complete the Self-Efficacy for Managing Chronic Disease Scale-6 (SEMCD-6) to assess self-efficacy in managing coronary artery disease. Scale scores range from 1 (minimum) to 10 (maximum), with higher scores indicating greater self-efficacy in managing chronic disease (i.e., a better outcome).
Self-efficacy for managing coronary artery disease | 30-day follow-up
  Participants will complete the Self-Efficacy for Managing Chronic Disease Scale-6 (SEMCD-6) to assess self-efficacy in managing coronary artery disease. Scale scores range from 6 (minimum) to 60 (maximum), with higher scores indicating greater self-efficacy in managing chronic disease (i.e., a better outcome).
Illness perceptions | 2-weeks/post-treatment
  Participants will complete the Brief Illness Perception Questionnaire (B-IPQ) as a measure of how threatening they perceive their coronary artery disease to be. Scale scores range from 0 (minimum) to 80 (maximum), with higher scores indicating more threatening illness perceptions (i.e., a worse outcome).
Illness perceptions | 30-day follow-up
  Participants will complete the Brief Illness Perception Questionnaire (B-IPQ) as a measure of how threatening they perceive their coronary artery disease to be. Scale scores range from 0 (minimum) to 80 (maximum), with higher scores indicating more threatening illness perceptions (i.e., a worse outcome).
Participant-reported depressive symptoms | 2-weeks/post-treatment
  The Patient Health Questionnaire-9 (PHQ-9) will be administered to assess depressive symptoms. Scale scores range from 0 (minimum) to 27 (maximum) with higher scores indicating elevated depressive symptoms (i.e., a worse outcome).
Participant-reported depressive symptoms | 30-day follow-up
  The Patient Health Questionnaire-9 (PHQ-9) will be administered to assess depressive symptoms. Scale scores range from 0 (minimum) to 27 (maximum) with higher scores indicating elevated depressive symptoms (i.e., a worse outcome).
Participant-reported anxiety symptoms | 2-weeks/post-treatment
  The Generalized Anxiety Disorder-7 (GAD-7) will be administered to assess anxious symptoms. Scale scores range from 0 (minimum) to 21 (maximum), with higher scores indicating elevated levels of anxiety symptoms (i.e., a worse outcome).
Participant-reported anxiety symptoms | 30-day follow-up
  The Generalized Anxiety Disorder-7 (GAD-7) will be administered to assess anxious symptoms. Scale scores range from 0 (minimum) to 21 (maximum), with higher scores indicating elevated levels of anxiety symptoms (i.e., a worse outcome).

SECONDARY OUTCOMES:
Participant-reported symptoms of demoralization | 2-weeks/post-treatment, 30-day follow-up
  Symptoms of demoralization will be measured using the Demoralization Scale-II (DS-II). Scale scores range from 0 (minimum) to 32 (maximum), with higher scores indicating more demoralization (i.e., a worse outcome).
Dietary patterns as measured using the brief dietary assessment and intervention tool: the Starting the Conversation (STC) questionnaire. | 2-weeks/post-treatment, 30-day follow-up
  Participants will report dietary patterns using the Starting the Conversation (STC) questionnaire. Scale scores range from 0 (minimum) to 16 (maximum) with lower scores indicating healthier dietary patterns (i.e., a better outcome).
Physical activity patterns | 2-weeks/post-treatment, 30-day follow-up
  The Global Physical Activity Questionnaire (GPAQ) will be administered to participants as a measure of physical activity behavior.
Number of cigarettes smoked per week over the past two weeks | 2-weeks/post-treatment, 30-day follow-up
  Participants who smoked a cigarette in the past month will complete a smoking questionnaire that assesses the number of cigarettes smoked per week over the past two weeks, motivation and readiness to quit smoking, in addition to interest in receiving smoking cessation referrals.
Confidence in resisting over-eating and unhealthy foods (i.e., Diet self-efficacy) | 2-weeks/post-treatment, 30-day follow-up
  Participant diet self-efficacy will be assessed with the scenario-based measure The Diet Self Efficacy Scale (DIET-SE). Scale scores range from 0 (minimum) to 44 (maximum), with higher scores indicating greater self-efficacy/confidence in dieting situations (i.e., a better outcome).
Confidence in exercising consistently (i.e., Exercise self-efficacy) | 2-weeks/post-treatment, 30-day follow-up
  Participant self-efficacy for exercise will be measured using the Exercise Confidence Survey (ECS). Scores range from 12 (minimum) to 60 (maximum), with higher scores indicating greater self-efficacy for exercise (i.e., a better outcome).

OTHER OUTCOMES:
Satisfaction with CLIMB intervention | 2-weeks/post-treatment (only for those who received the intervention)
  Participants will complete a satisfaction survey regarding their participation in the CLIMB intervention.
Program development questionnaire | 2-weeks/post-treatment (only for those who received the intervention)
  Participants will complete a program development questionnaire regarding their participation in the CLIMB intervention to inform further development of the intervention.
CLIMB Intervention Acceptability: Would participants recommend this intervention to other patients with coronary artery disease? | 2-weeks/post-treatment (only for those who received the intervention)
  Acceptability of the intervention will be assessed with the Yes/No question: "Would you recommend this intervention to other patients with coronary artery disease?" At least 80% need to respond "Yes" for the treatment to be considered acceptable.
Percentage of referred and eligible patients agreeing to participate (Feasibility Assessment) | Through study completion: anticipated 1 year
  The program will only be considered feasible if at least 60% of referred and eligible patients agree to participate.
Percentage of participants completing CLIMB intervention through 30-day follow-up (Feasibility Assessment) | Through study completion: anticipated 1 year
  The study will only be considered feasible if at least 75% of the consented IG participants complete the study intervention and outcome measurements through the 30-day follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea H. Wiener, MS, Principal Investigator — University of Central Florida
Locations (1):
- UCF Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No